CLINICAL TRIAL: NCT03891043
Title: Oral Supplementation With Selenium in Patients With Mild Thyroid Orbitopathy to Reduce Its
Brief Title: Oral Supplementation With Selenium in Patients With Mild Thyroid Orbitopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CI-043-2015
Record Dates: First submitted 2019-03-15; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2018-09

CONDITIONS: Thyroid Orbitopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A, Placebo group (Placebo Comparator): Placebo consisted in a pill of 100 micrograms of starch, to be taken twice a day.
  Interventions: Other: Placebo
- Group B, Selenium group (Experimental): Selenium consisted in a pill of 100 micrograms, to be taken twice a day.
  Interventions: Dietary Supplement: Selenium

INTERVENTIONS:
Dietary Supplement: Selenium — A 100 micrograms of Selenium was given to be taken twice a day.
  Arms: Group B, Selenium group
Other: Placebo — Placebo pill of 100 micrograms of starch was given to be taken twice a day.
  Arms: Group A, Placebo group

SUMMARY:
Background: The activity of thyroid orbitopathy can be evaluated with CAS (Clinical Activity Score) based on 7 inflammatory signs. Selenium acts as an oxide-reducing agent in thioredoxin-reductase, and as an anti-inflammatory agent by reducing the hydroxy peroxide intermediates on the cyclo-oxygenase pathways. Increased oxidative stress has been observed in Graves' disease and therefore, by incorporating an antioxidant such as selenium in patients with mild thyroid ophthalmopathy, inflammatory activity could be reduced or inactivated.

General Objective: To determine the clinical differences between patients with mild thyroid orbitopathy who were administered oral supplementation with selenium and patients who were administered oral placebo.

DETAILED DESCRIPTION:
This is a simple controlled clinical trial. In which 66 eyes of 33 patients were studied. Fifteen patients were assigned to the placebo group and 18 to the Selenium group. We randomized into two groups the patients with mild clinical activity according to CAS score. Group A took placebo pills twice a day which consisted in 100µg of starch, and Group B took a pill of Selenium 100 µg twice a day. All the subjects tool the pills during six months. Patients of both groups where examined and evaluated with CAS score before and after the first, third and sixth month of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active mild thyroid orbitopathy according to CAS scale.
* Older than 18 years of age.

Exclusion Criteria:

* Patients with mild thyroid orbitopathy undergoing treatment with corticosteroids.
* Active smokers
* Patients allergic to Selenium
* Follow-up shorter than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Clinical Activity Score (CAS) | 6 months after treatment
  Clinical Activity Score (CAS) scale consists of 7 measurements used to evaluate clinical activity of thyroid orbitopathy:
  1. Spontaneus orbital pain
  2. Gaze evoked orbital pain
  3. Conjunctival redness that is considered to be due to active GO
  4. Eyelid erythema
  5. Chemosis
  6. Eyelid swelling that is considered to be due to active GO
  7. Inflammation of plica or caruncle